CLINICAL TRIAL: NCT02355197
Title: Physiological Effects of Gestational Diabetes on the Placenta and Neonatal Outcome; Role of Antioxidant Administration
Brief Title: Antioxidants in Gestational Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124
Record Dates: First submitted 2015-01-26; First posted 2015-02-04 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Gestational Diabetes Mellitus
Keywords: antioxidants; Gestational diabetes mellitus; oxidative stress
MeSH Terms: conditions — Diabetes, Gestational | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antioxidant (Active Comparator): 1 gram L-ascorbic acid (vitamin C capsule) orally once per day from the time of diagnosis until the time of delivery in addition to treatment for gestational diabetes mellitus in the form of diet and insulin
  Interventions: Drug: L-ascorbic acid
- control (No Intervention): Only treatment for gestational diabetes mellitus in the form of diet and insulin

INTERVENTIONS:
Drug: L-ascorbic acid — 1 gram L-ascorbic acid (vitamin C …..) per day from the time of diagnosis until the time of delivery
  Other Names: vitamin C
  Arms: antioxidant

SUMMARY:
Fasting and two hours postprandial blood sugar were done to all cases between 28 and 32 weeks and high blood sugar levels were found so Cases were controlled by both diet and insulin.

The 200 pregnant women with Gestational diabetes mellitus were randomized using automated web based randomization system into 2 groups, Group1 received 1 gram L-ascorbic acid (vitamin C )per day from the time of diagnosis until the time of delivery in addition to routine treatment of diabetes (diet & insulin). Group2 received only the treatment of diabetes

DETAILED DESCRIPTION:
The 200 pregnant women with Gestational diabetes mellitus were randomized using automated web based randomization system into 2 groups, Group1 received 1 gram L-ascorbic acid oral once daily (vitamin C )per day from the time of diagnosis until the time of delivery in addition to routine treatment of diabetes (diet & insulin). Group2 received only the treatment of diabetes (diet and insulin

ELIGIBILITY:
Inclusion Criteria:

* Women with the diagnosis of GDM

Exclusion Criteria:

* Women with multiple pregnancies
* Chronic medical disorders e.g. anemia
* Hypertension
* Liver disease or renal disease
* Those with obstetric problems other than GDM (e.g. pre-eclampsia & antepartum hemorrhage) or smokers and women with preexisting type I or II diabetes mellitus were excluded from our study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
neonatal outcome assessed by neonatal ICU admission | 1 week after delivery

SECONDARY OUTCOMES:
oxidative stress parameters: non enzymatic and enzymatic oxidative stress parameters in placental tissue homogenates in women with GDM named glutathione ,malondialdahyde,superoxide dismutase ,catalase and glutathione peroxidase | 9 months of pregnancy
oxidative stress parameters: non enzymatic and enzymatic oxidative stress parameters in maternal blood plasma/lysate in women with GDM named glutathione,superoxide dismutase ,catalase and glutathione peroxidase | 9 months of pregnancy
oxidative stress parameters: non enzymatic and enzymatic oxidative stress parameters in neonatal blood in women with GDM named malondialdahyde and superoxide dismutase | 9 months of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt